CLINICAL TRIAL: NCT02996669
Title: Autism Biomarker Consortium for Clinical Trials
Acronym: ABC-CT
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Boston Children's Hospital (Other); Duke University (Other); University of California, Los Angeles (Other); University of Washington (Other); Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1509016477; U01FD006888 (FDA); U19MH108206 (NIH)
Record Dates: First submitted 2015-10-21; First posted 2016-12-19 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: During Screening Visits, the Autism Diagnostic Observational Schedule (ADOS) will be administered to confirm diagnosis. Criteria for group inclusion is: diagnosis of Autism Spectrum Disorder based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-G), and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
- Typical Development: Typically Developing (TD) participants from each site will be roughly matched by age and sex to the ASD group.

SUMMARY:
This is a multicenter longitudinal study that aims to identify, develop and validate a set of measures that can be used as stratification biomarkers and/or sensitive and reliable objective measures of social impairment in autism spectrum disorders (ASD) that could serve as markers of long term clinical outcome. The main study will include 275 individuals: 200 ASD subjects between 6-11 years old, and 75 TD subjects roughly matched by age and sex to the ASD group.

DETAILED DESCRIPTION:
The specified aims of this study are to accelerate the development of effective treatments for social impairment in ASD by validating outcome measures that will be sensitive and reliable assessments of response to treatment and electroencephalography (EEG) and eye-tracking (ET) biomarkers. These hypothesized outcomes could then be used to reduce the heterogeneity of samples via stratification, could possibly indicate early efficacy, and/or demonstrate target engagement. The consortium will conduct a naturalistic, longitudinal study of preschool and school-aged (6-11 years) children with ASD and typical development (TD) with intelligence quotient(s) (IQ) ranging from 50-150. Children will be assessed across three time points (Baseline, 6 weeks and 24 weeks) using clinician, caregiver and lab-based (LB) measures of social impairment, along with a battery of conceptually related EEG and ET tasks and independent ratings of clinical status.

ELIGIBILITY:
Inclusion Criteria:

For All Subjects:

* Males and Females Age 6 - 11 (<11:5 at timepoint #1 unless all study procedures will be completed before the participant turns 12.0 and prior approval by the Principal Investigator is obtained).
* Written parental consent obtained prior to any study procedures.
* Participant and parent/guardian must be English speaking.

For TD Participants:

• IQ 80-150 as assessed by the Differential Ability Scales (DAS)- 2nd Edition

For ASD Participants:

* Diagnosis of ASD based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-2), and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
* IQ 60-150 as assessed by the Differential Ability Scales (DAS)- 2nd Edition
* If parents are biological, a minimum of the child and one parent (if accompanying the child at study visits) will be required to participate in the blood draw procedure. It is preferred that the child and both biological parents participate in the blood draw procedure, but the inability to obtain blood samples from trios will not be exclusionary.

Exclusion Criteria:

For All Subjects:

* Known genetic or neurological syndrome with established link to autism (in addition to ASD for ASD participants), but not events in which the link to ASD is less well known/established (e.g., 16p11.2 CNVs, CHD8 mutations, Trisomy 21, 22q deletion syndrome)
* History of epilepsy or seizure disorder (except for history of simple febrile seizures or if the child is seizure free (regardless of seizure type) for the past year).
* Motor or sensory impairment that would interfere with the valid completion of study measures including significant hearing or vision impairment not correctable by a hearing aid or glasses/contact lenses. Children who wear bifocal or progressive lenses are not eligible.
* Medication is not exclusionary. Children taking neurological or psychiatric medications, including anti epileptics and psychopharmacological agents, must be stable on the medication and dose for 8 weeks prior to T1D1.
* History of significant prenatal/perinatal/birth injury (birth <36 weeks AND weight <2000 grams (approximately 4.5lbs)).
* History of neonatal brain damage. (e.g., with diagnoses hypoxic or ischemic event)
* Any other factor that the investigator feels would make assessment or measurement performance invalid.

For ASD Participants:

• Any known environmental circumstances that is likely to account for the picture of autism in the proband (severe nutritional or psychological deprivation etc.)

For TDs Participants:

* Known historical diagnosis of ASD or a sibling with ASD.
* Active psychiatric disorder (depression, anxiety, ADHD, etc.) and/or any current treatment (medication or other treatment) for a psychiatric condition. Participants will be screened using the Child/Adolescent Symptom Inventory (CASI-5). Due to the measurements sensitivity, any score in the clinical range will be reviewed by research staff for determination of eligibility.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 children with an autism spectrum disorder between 6-11 years old, and 75 typically developing children
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2016-10; Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
NEPSY-II | Baseline
  NEPSY-II - Memory for Faces Subtest (administered to all ages): The NEPSY-II Memory for Faces subtest entails viewing a series of faces and having the child identify the sex of each face. The child is then shown three faces at a time and required to identify the previously seen face.
NEPSY-II | 6 weeks
  NEPSY-II - Memory for Faces Subtest (administered to all ages): The NEPSY-II Memory for Faces subtest entails viewing a series of faces and having the child identify the sex of each face. The child is then shown three faces at a time and required to identify the previously seen face.
NEPSY-II | 24 weeks
  NEPSY-II - Memory for Faces Subtest (administered to all ages): The NEPSY-II Memory for Faces subtest entails viewing a series of faces and having the child identify the sex of each face. The child is then shown three faces at a time and required to identify the previously seen face.
Video Tracking | Baseline
  Video tracking of social behavior is an observational method involving automated tracking of children's movements using the Noldus EthoVision Computerized tracking system. Using computer vision, video recordings of children's movements assess proximity-seeking/approach behaviors. During one six-minute free-play session in the laboratory, children's movements will be recorded from a ceiling-mounted camera and two side cameras while a parent sits in a corner of the room. Software automatically tracks the child (via the ceiling mounted camera) as the child plays with a standardized set of toys and interacts with the parent, and computes the percentage of session spent near the parentlatency to approach the parent, percentage of time spent in the periphery and latency to approach the periphery. A subset of side camera recordings will be manually coded by reliable coders for social engagement behaviors to validate the automatically generated movement behaviors calculated by EthoVision.
Video Tracking | 6 weeks
  Video tracking of social behavior is an observational method involving automated tracking of children's movements using the Noldus EthoVision Computerized tracking system. Using computer vision, video recordings of children's movements assess proximity-seeking/approach behaviors. During one six-minute free-play session in the laboratory, children's movements will be recorded from a ceiling-mounted camera and two side cameras while a parent sits in a corner of the room. Software automatically tracks the child (via the ceiling mounted camera) as the child plays with a standardized set of toys and interacts with the parent, and computes the percentage of session spent near the parentlatency to approach the parent, percentage of time spent in the periphery and latency to approach the periphery. A subset of side camera recordings will be manually coded by reliable coders for social engagement behaviors to validate the automatically generated movement behaviors calculated by EthoVision.
Video Tracking | 24 weeks
  Video tracking of social behavior is an observational method involving automated tracking of children's movements using the Noldus EthoVision Computerized tracking system. Using computer vision, video recordings of children's movements assess proximity-seeking/approach behaviors. During one six-minute free-play session in the laboratory, children's movements will be recorded from a ceiling-mounted camera and two side cameras while a parent sits in a corner of the room. Software automatically tracks the child (via the ceiling mounted camera) as the child plays with a standardized set of toys and interacts with the parent, and computes the percentage of session spent near the parentlatency to approach the parent, percentage of time spent in the periphery and latency to approach the periphery. A subset of side camera recordings will be manually coded by reliable coders for social engagement behaviors to validate the automatically generated movement behaviors calculated by EthoVision.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) | Baseline, 6 weeks and 24 weeks
  The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors of children and adults with neurodevelopmetnal disorder at home, in residential facilities, ICFs/MR, and work training centers. It is also useful for classifying problem behaviors of children and adolescents with neurodevelopmetnal disorder in educational settings, residential and community-based facilities, and developmental centers.
  Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985; 89(5):485-491.
Autism Impact Measure (AIM) Frequency | Baseline, 6 weeks and 24 weeks
  The Autism Impact Measure (AIM) uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact). PMID: 23748386.
Autism Impact Measure (AIM) Impact | Baseline, 6 weeks and 24 weeks
  The Autism Impact Measure (AIM) uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact). PMID: 23748386.
Child and Adolescent Symptom Inventory 5 (CASI-5) | Baseline, 6 weeks and 24 weeks
  The Child & Adolescent Symptom Inventory-5 (CASI-5) is a behavior rating scale for DSM-5-defined emotional and behavioral disorders in youths between 5 and 18 years old.
PDD Behavior Inventory (PDD-BI) | Baseline, 6 weeks and 24 weeks
  The PDD-BI is an assessment tool for children on the autism spectrum. PDDBI profiles can provide guidance to clinicians regarding the child's problems as perceived by the informants, how a particular child compares to most children their age with ASD, and the skills and abilities of the child.
  Cohen, I. L. (2003). Criterion-related validity of the PDD Behavior Inventory. Journal of Autism and Developmental Disorders, 33, 47-53.
Social Responsiveness Scale 2 (SRS-2) Total Score | Baseline, 6 weeks and 24 weeks
  The Social Responsiveness Scale 2 (SRS-2) is completed in just 15 to 20 minutes and identifies social impairment associated with autism spectrum disorders (ASDs) and quantifies its severity.
Cognitive Assessment | Baseline and 24 weeks
  Differential Ability Scales - Second Edition; DAS-II (Elliott C, 2007): The DAS-II is a clinical instrument designed to assess cognitive ability include variables such as verbal cluster, spatial cluster, nonverbal cluster, special nonverbal composite and GCA. The overall score will be used.
Resting State EEG | Baseline, 6 weeks and 24 weeks
  Resting State EEG (Eyes Open) provides a reference for the event-related EEG measures and a baseline biomarker of EEG spectral power across frequencies, neurofunctional connectivity and coherence, and hemispheric asymmetry and will always be done prior to the other EEG paradigms. Participants will be presented with non-social, abstract moving videos in random order.
Faces EEG | Baseline, 6 weeks and 24 weeks
  Faces processing is a foundation for social perception and attention and serves as a promising and robust biomarker of social impairment in ASD and a potential index of subgroup differences. As the primary non-resting paradigm, the FACES task will always be administered second in the EEG protocol. Participants will be presented with a series of upright and inverted faces, as well as upright houses (as a contrast non-face stimulus).
Visual Evoked Potentials (VEPs) EEG | Baseline, 6 weeks and 24 weeks
  Visual Evoked Potentials (VEPs) index low-level visual processing and reflect the functional integrity of the visual pathway. VEPs reflect excitatory (glutamatergic) and inhibitory (GABAergic) activity and may index subgroups of ASD with low-level visual impairments. VEPs also serve as a control for assessment of higher-order activity in social visual paradigms. Subjects will be presented with black and white checkerboards that reverse phase at a defined interval. The order of the VEP and Biomotion paradigms will be counterbalanced.
Biological Motion EEG | Baseline, 6 weeks and 24 weeks
  Biological Motion processed by specific neural circuitry, which has demonstrated to exhibit reduced sensitivity in ASD. Point light displays (PLDs) of a human walking versus scrambled motion will be presented randomly. The order of the VEP and Biomotion paradigms will be counterbalanced.
Eye-tracking (ET) Biological Motion Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Biological Motion Task is measured after short central fixation, children will be presented with Point Light Displays (PLDs) indicating target biological motion and a scrambled or a rotating perceptual control.
Eye-tracking (ET) Activity Monitoring Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Activity Monitoring Task is measured following central fixation. Children will be presented with multiple activity monitoring trails depicting two actresses engaging in a controlled joint activity such as assembling a puzzle.
Eye-tracking (ET) Interactive Social Task (IST) | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Interactive Social Task (IST) is taps similar constructs as the activity monitoring task in a more naturalistic, dynamic, and complex context. Following a central fixation, children will be presented with interactive social trails in which two children engage in a natural interactive play session.
Eye-tracking (ET) Pupillary Light Reflex Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Pupillary Light Reflex (PLR) Task is measured following a stimuli that consist of a central fixation point on a black background that flashes white for 133 milliseconds. The constriction of the pupil in response to a bright flash indexes function of the parasympathetic nervous system.
Eye-tracking (ET) Visual Search/Static Social Scenes Task | Baseline, 6 weeks and 24 weeks
  ET Paradigms will be administered in counterbalanced blocks, one on each day of each screening or study visits. Both blocks will include all the tasks but in different orders. The length of individual paradigms ranges from 1 to 8.5 mins.
  Color images depicting 12 different female faces with direct gaze and the same faces with averted gaze will be presented. Twelve different exemplars from each of five categories (alarm clocks, mobile phones, birds, cars, and shoes) will be used as distracters. Twelve different slides will each contain six images (one face and five distracters, one from each category) placed at an equal distance from the center of the screen. Each slide contains a different set of six images, each image being shown only once in the experiment. This measure examines scanning patterns towards arrays of objects, synthetic stimuli, and faces as well as towards more complex naturalistic (static) scenes. This task examines complex scene processing and attentional select

CONTACTS AND LOCATIONS:
Overall Officials: James McPartland, PhD, Principal Investigator — Yale University Child Study Center
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Faja S, Sabatos-DeVito M, Sridhar A, Kuhn JL, Nikolaeva JI, Sugar CA, Webb SJ, Bernier RA, Sikich L, Hellemann G, Senturk D, Naples AJ, Shic F, Levin AR, Seow HA, Dziura JD, Jeste SS, Chawarska K, Nelson CA 3rd, Dawson G, McPartland JC; Autism Biomarkers Consortium for Clinical Trials. Evaluation of clinical assessments of social abilities for use in autism clinical trials by the autism biomarkers consortium for clinical trials. Autism Res. 2023 May;16(5):981-996. doi: 10.1002/aur.2905. Epub 2023 Mar 16. PMID 36929131
- [Derived] Shic F, Naples AJ, Barney EC, Chang SA, Li B, McAllister T, Kim M, Dommer KJ, Hasselmo S, Atyabi A, Wang Q, Helleman G, Levin AR, Seow H, Bernier R, Charwaska K, Dawson G, Dziura J, Faja S, Jeste SS, Johnson SP, Murias M, Nelson CA, Sabatos-DeVito M, Senturk D, Sugar CA, Webb SJ, McPartland JC. The autism biomarkers consortium for clinical trials: evaluation of a battery of candidate eye-tracking biomarkers for use in autism clinical trials. Mol Autism. 2022 Mar 21;13(1):15. doi: 10.1186/s13229-021-00482-2. PMID 35313957